CLINICAL TRIAL: NCT00525564
Title: Effects of Salmeterol on Walking Capacity in Patients With COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SMS106875
Record Dates: First submitted 2007-09-04; First posted 2007-09-06 (Estimated); Last update posted 2007-09-06 (Estimated); Status verified 2007-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease (COPD); Exercise; Endurance shuttle walking test; Bronchodilation; Salmeterol
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Salmeterol Xinafoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Placebo Comparator): Placebo diskus
  Interventions: Drug: Placebo
- B (Active Comparator): Salmeterol diskus powder
  Interventions: Drug: Salmeterol diskus inhalation powder

INTERVENTIONS:
Drug: Placebo — Placebo diskus inhalation powder
  Arms: A
Drug: Salmeterol diskus inhalation powder — 50 micrograms twice a day
  Other Names: Serevent
  Arms: B

SUMMARY:
This study was designed to test the following hypothesis:

The acute changes in exercise tolerance during the endurance shuttle walk will be greater with salmeterol compared to placebo in patients with chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
Background: Little is known about the responsiveness of the endurance shuttle walking test (ESWT) to pharmacotherapy in patients with chronic obstructive pulmonary disease (COPD). This exercise testing modality needs to be further investigated because of its relevance for activity of daily living.

Objective: To evaluate, in patients with COPD, the responsiveness of the ESWT to detect improvement in walking performance after single dose of salmeterol.

Methods: In a randomised, double-blind, placebo-controlled, crossover study, 20 patients with COPD will perform, on two separate days, an ESWT at 80% of peak capacity, 2 hours after inhaling either a placebo or 50µg of salmeterol. Cardiorespiratory parameters will be monitored breath-by-breath during each walking test with a portable telemetric gas analyzer (Oxycom Mobile, Jaeger, Germany). Inspiratory capacities and Borg ratings for dyspnea were obtained every other minute throughout the tests.

Planned analysis. The main outcome will be endurance time. This variable will be compared between the two treatment arms using a paired t test. The time course of the cardiorespiratory parameters and dyspnea over time will be compared between the two exercise modalities. Comparisons will be done using a repeated measure design (ANOVA). Significance level will be set at a p value of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* age > 50 years
* smoking history > 10 packs/year
* FEV1 < 70% of predicted and FEV1/FVC < 70%.

Exclusion Criteria:

* respiratory exacerbation within the 2 months preceding the study
* history of asthma
* significant O2 desaturation (SaO2 < 85%) at rest or during exercise
* presence of another pathology that could influence exercise tolerance.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-05; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Endurance time during an endurance shuttle walk | acute response (2.5 hours) following the administration of the active and comparison drug

SECONDARY OUTCOMES:
Dyspnea during endurance shuttle walk | acute response following the administration of the study medication
cardio-respiratory responses during an endurance shutlle walk | acute response following the administration of the study medication

CONTACTS AND LOCATIONS:
Overall Officials: François Maltais, MD, Principal Investigator — Laval University
Locations (1):
- Hôpital Laval, Québec, Quebec, Canada